CLINICAL TRIAL: NCT05281822
Title: Sivas Cumhuriyet University, Faculty of Health Sciences
Brief Title: The Stress Management Training Provided to Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Assoc. Prof. Dr, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SIVAS 01
Record Dates: First submitted 2022-03-03; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Obese Women; Stress; Training
Keywords: women; obesity; stress; stress management training; eating attitude
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The BMI (kg/m2) was calculated by measuring the height and weight of the women in the experimental groups. Then, the women in the experimental group were provided with stress management training to help cope with stress conditions, how to use positive coping in conditions in case of stress and tension. In terms of the reliability of the training, each woman was interviewed face-to-face, which lasted for 30-40 minutes.
  Interventions: Other: The stress management training

INTERVENTIONS:
Other: The stress management training — The women in the experimental group were provided with stress management training to help cope with stress conditions how to use positive coping in conditions in case of stress and tension.

SUMMARY:
Introduction: Obesity, which is an important public healthcare issue, can affect women's physical, mental, social health, stress level, and coping negatively.

Aim: The present study was conducted to determine the effects of stress management training provided to obese women on eating attitudes, stress, and coping with stress.

DETAILED DESCRIPTION:
Methods: The sampling of the randomized controlled experimental study based on the pre-test and post-test model consisted of 70 women (experimental = 35; control = 35) with a Body Mass Index ≥30, who applied to a Community Healthcare Center Obesity Unit in primary care in Turkey. The data were collected by using Personal Information Form, Perceived Stress Scale, Stress Coping Styles Scale, Dutch Eating Behavior Questionnaire, and height-weight measurements.

ELIGIBILITY:
Inclusion Criteria:

* Women who lived in the city center,
* Body Mass Index ≥30,
* Having no perception and communication problems and being able to answer questions,
* Women who volunteered to participate in the study

Exclusion Criteria:

* Being a man
* Non-obese women and those with a body mass index below 30
* Those with communication problems
* Those who do not live in the city center

Ages: 23 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 10 months
  The scale consisted of 10 items, scored between 1-5 and the total score is calculated between 10-50. As the score increases, the stress level also increases.
Styles of Coping with Stress Inventory | 10 months
  The scale, which consists of a total of 30 items, is scored between 0-3. The scores of each sub-dimension are calculated separately, the total score is not calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sukran Ertekin Pinar, Principal Investigator — Cumhuriyet University
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No